CLINICAL TRIAL: NCT02498132
Title: Development and Testing of a Behavioral Activation Mobile Therapy for Elevated Depressive Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: MOUNTAINPASS TECHNOLOGY, LLC (Unknown); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Joe Smith, Director - HRPP (C. Lejuez is no longer at UMD), University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R41MH108219-01 (NIH)
Record Dates: First submitted 2015-07-07; First posted 2015-07-15 (Estimated); Results first posted 2022-02-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: Mobile Technologies
MeSH Terms: conditions — Depression | interventions — Therapeutics

ARMS (3):
- Behavioral Activation (Experimental): Behavioral Activation will be administered via Moodivate will mirror the core BA components outlined above. Moodivate will also be modified for a mobile environment in key ways, with the most salient being: 1) Elimination of the need for a therapist: By eliminating the need for a therapist, we will be able to reach a broad patient/consumer base that may not utilize traditional therapy resources and will combat the primary barrier to PCPs recommending psychotherapy to their patients with elevated depressive symptoms and 2) Elimination of paper forms: By eliminating paper forms, we will increase the sensitivity of BA to motivational and organizational deficits frequently observed in patients with elevated depressive symptoms while also increasing treatment fidelity by prompting the patient to complete activities at scheduled times and giving the patient reinforcement for completing activities.
  Interventions: Other: Behavioral Activation
- Cognitive Based Therapy (Active Comparator): Moodkit will be used to administer cognitive based therapy which is commonly compared to behavioral activation.
  Interventions: Other: Cognitvie Based Therapy
- Treatment as Usual (Active Comparator): TAU will be provided to individuals. These subject will be provided with therapy but will not utilize a mobile application.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Behavioral Activation — BA is based in behavioral principles of depression that suggest that depression is caused by a lack of reinforcement in the environment for positive, non-depressed behaviors. As such, the goal of BA is to help the patient reengage in positive, non-depressed activities. In clinical trials, BA as a treatment component has been consistently superior to no treatment and treatment as usual control groups, and a large body of research has found that BA is either equally or more effective than CBT, CT, and antidepressant medications (Cuijpers, Van Straten, & Warmerdam, 2007; Dimidjian et al., 2006; Jacobson et al., 1996).
  Arms: Behavioral Activation
Other: Cognitvie Based Therapy — CBT explores patterns of thinking that lead to self-destructive actions and the beliefs that direct these thoughts, people with mental illness can modify their patterns of thinking to improve coping
  Arms: Cognitive Based Therapy
Other: Treatment as Usual — Individuals will be provided with one on one therapy sessions
  Arms: Treatment as Usual

SUMMARY:
Elevated depressive symptomatology is a widespread public health concern and individuals with elevated depressive symptoms most frequently report such symptoms to primary care physicians (PCPs). PCPs have few evidence-based resources beyond antidepressant medication for treating elevated depressive symptoms, which results in negative outcomes for their depressed patients. Mobile technologies offer an ideal strategy to meet widespread treatment needs. The purpose of the proposed project is to\ customize Behavioral Activation (BA), a straightforward, empirically supported treatment for elevated depressive symptoms, for a mobile format (Moodivate) in order to address the currently unmet needs of PCPs and their patients with elevated depressive symptoms.

DETAILED DESCRIPTION:
Depressive symptoms are associated with heightened risk of developing major depressive disorder (MDD), significant public health costs, and mortality rates equal to MDD . Individuals experiencing impairment due to depressive symptomatology most frequently report their depressive symptoms to a primary care physician . Despite conflicting data regarding efficacy, PCPs typically prescribe antidepressant medication for the treatment of subthreshold depression and have few other resources at their disposal . The current lack of evidence-based resources available to PCPs for treating depressive symptoms results in a number of negative outcomes for patients including: 1) the majority not receiving appropriate treatment , 2) a decreased likelihood of reporting depressive symptoms again in the future , and 3) heightened mortality risk. As the most likely initial contact for patients with elevated depressive symptoms, PCPs are in a unique position to provide interventions for depression .

Mobile technologies offer an ideal strategy to meet widespread treatment needs. Mobile technologies broadly, and mobile phones more specifically, have dramatically increased in both affordability and ubiquity, with current estimates suggesting that there are over 3.2 billion unique mobile users worldwide . Moreover, the vast majority of physicians report using mobile apps in their clinical practice . Despite these factors supporting the use of mobile apps in clinical practice, there are currently no mobile apps for depressive symptoms available to PCPs that are both evidence-based and simple enough to be recommended to their patients.

One treatment that is particularly amenable to a mobile platform and to referral by PCPs is Behavioral Activation. Across studies, BA is effective for reducing depressive symptoms among individuals with subthreshold depression as well as individuals with MDD and meets the criteria to be established as an empirically support treatment . Moreover, numerous research studies support the superiority of BA as a treatment component to competitor treatments, including Cognitive Behavioral Therapy (CBT) and Cognitive Therapy (CT). The cornerstone of BA is regular self-monitoring to 1) examine already occurring daily activities and 2) facilitate incorporation of new activities consistent with individualized values and goals across life areas. Empirical evidence indicates that mobile customization of BA would work as intended to facilitate reduction of depressive symptomatology, while also addressing the unmet need for evidence-based and easily disseminable resources for use by PCPs with their patients with depressive symptomatology. Moreover, as BA has an evidence-base for smoking cessation, a mobile customization of BA may also hold promise for promoting smoking cessation.

With STTR funding from NIMH, our team is currently completing the development of a self-help BA mobile application named Moodivate for referral by PCPs to their patients with elevated depressive symptoms. App development will be complete by March, 2016 in preparation for a small clinical trial at MUSC. The closest competitor apps for Moodivate are Cognitive Behavioral Therapy (CBT)-based mobile applications. The most popular CBT-based mobile applications include iCouch CBT, Live Happy, MoodPanda, and MoodKit. Of this group of CBT-based mobile applications, MoodKit most closely adheres to standard CBT. As clinical trials of standard BATD frequently compare BATD to CBT, an appropriate analogue of this line of work is to compare Moodivate, a BATD based mobile app, to MoodKit, a CBT based mobile app. Although MoodKit appears to adhere to CBT, no clinical trials to date have been completed examining utilization of MoodKit among individuals with elevated depressive symptoms or among individuals referred by a PCP.

In the current study, we will conduct a small-scale randomized clinical trial with 60 adults with elevated depressive symptoms (Beck Depression Inventory-II (BDI-II) > 14; above the "minimal depression" range on the measure) referred from physicians in the Department of Family Medicine (Drs. Vanessa Diaz and Marty Player) at MUSC. Participants will be randomized to one of three conditions: 1) Moodivate, 2) a Cognitive Behavioral Therapy-based mobile application (MoodKit), or 3) Treatment As Usual (TAU). The purpose of this step is to examine Moodivate treatment feasibility, acceptability, adherence, and change in depressive symptoms associated with Moodivate as compared to MoodKit and TAU. Considering that BA also has an evidence base for smoking cessation, within this group of 60 participants, we plan to recruit 10 participants who are current smokers who will receive Moodivate. Although this will be a small sample of smokers receiving the BA mobile therapy, we believe collecting pilot data examining utilization of Moodivate among a group of smokers will provide valuable insight into the feasibility of utilizing a BA mobile app to promote smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

Participants will be screened by phone. Inclusion criteria:

Participants must:

1. be between the ages of 18 and 65,
2. report current elevated depressive symptoms, and
3. currently own an iOS-compatible mobile phone.

Exclusion Criteria:

Participants will be excluded if they:

1. are currently receiving psychotherapy or psychotropic medication,
2. plan to seek psychotherapy within the next 3 months (score > 5 on a self-report 1-10 scale of likelihood to seek treatment),
3. endorse current suicidal ideation defined as either

   1. a response of "I would like to kill myself" or "I would kill myself if I had the chance" on the suicidal thoughts or wishes item of the BDI-II or
   2. an indication of past month suicidal ideation on the MDD module of the SCID-IV (see Protection of Human Subjects for additional details), or
4. meet current diagnostic criteria for MDD; although BA has been used to treat MDD, Moodivate is targeted specifically to elevated symptoms, not major depressive episodes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Lejuez, Ph.D., Principal Investigator — University of Maryland, College Park; Jennifer Dahne, MS, Study Chair — University of Maryland, College Park

REFERENCES:
- [Background] Kubik MY, Lytle LA, Birnbaum AS, Murray DM, Perry CL. Prevalence and correlates of depressive symptoms in young adolescents. Am J Health Behav. 2003 Sep-Oct;27(5):546-53. doi: 10.5993/ajhb.27.5.6. PMID 14521250
- [Background] Cuijpers P, Vogelzangs N, Twisk J, Kleiboer A, Li J, Penninx BW. Differential mortality rates in major and subthreshold depression: meta-analysis of studies that measured both. Br J Psychiatry. 2013 Jan;202(1):22-7. doi: 10.1192/bjp.bp.112.112169. PMID 23284149
- [Background] Mitchell AJ, Vaze A, Rao S. Clinical diagnosis of depression in primary care: a meta-analysis. Lancet. 2009 Aug 22;374(9690):609-19. doi: 10.1016/S0140-6736(09)60879-5. Epub 2009 Jul 27. PMID 19640579
- [Background] Kessler RC, Demler O, Frank RG, Olfson M, Pincus HA, Walters EE, Wang P, Wells KB, Zaslavsky AM. Prevalence and treatment of mental disorders, 1990 to 2003. N Engl J Med. 2005 Jun 16;352(24):2515-23. doi: 10.1056/NEJMsa043266. PMID 15958807
- [Background] Bell RA, Franks P, Duberstein PR, Epstein RM, Feldman MD, Fernandez y Garcia E, Kravitz RL. Suffering in silence: reasons for not disclosing depression in primary care. Ann Fam Med. 2011 Sep-Oct;9(5):439-46. doi: 10.1370/afm.1277. PMID 21911763
- [Background] Cuijpers P, de Graaf R, van Dorsselaer S. Minor depression: risk profiles, functional disability, health care use and risk of developing major depression. J Affect Disord. 2004 Apr;79(1-3):71-9. doi: 10.1016/S0165-0327(02)00348-8. PMID 15023482
- [Background] McDowell AK, Lineberry TW, Bostwick JM. Practical suicide-risk management for the busy primary care physician. Mayo Clin Proc. 2011 Aug;86(8):792-800. doi: 10.4065/mcp.2011.0076. Epub 2011 Jun 27. PMID 21709131
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Gawrysiak, M., Nicholas, C., & Hopko, D. R. (2009). Behavioral activation for moderately depressed university students: Randomized controlled trial. Journal of Counseling Psychology, 56(3), 468-475.
- [Background] Hopko DR, Lejuez CW, LePage JP, Hopko SD, McNeil DW. A brief behavioral activation treatment for depression. A randomized pilot trial within an inpatient psychiatric hospital. Behav Modif. 2003 Sep;27(4):458-69. doi: 10.1177/0145445503255489. PMID 12971122
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). Beck Depression Inventory-II (BDI-II). San Antonio, TX: Psychological Corporation.
- [Background] McNair, D. M., Lorr, M., & Droppleman, L. F. (1971). Manual for the profile of mood states (POMS). San Diego, CA: Educational and Industrial Testing Services.
- [Background] First, M., Spitzer, R., Gibbon, M., & Williams, J. (2002). Structured Clinical Interview for DSM-IV Axis IDdisorders: Research Version: Non-patient Edition (SCID-I/NP). New York, NY: Biometrics Research, New York State Psychiatric Insititute.
- [Background] Cuijpers P, van Straten A, Warmerdam L. Behavioral activation treatments of depression: a meta-analysis. Clin Psychol Rev. 2007 Apr;27(3):318-26. doi: 10.1016/j.cpr.2006.11.001. Epub 2006 Dec 19. PMID 17184887
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Jacobson NS, Dobson KS, Truax PA, Addis ME, Koerner K, Gollan JK, Gortner E, Prince SE. A component analysis of cognitive-behavioral treatment for depression. J Consult Clin Psychol. 1996 Apr;64(2):295-304. doi: 10.1037//0022-006x.64.2.295. PMID 8871414

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Activation: Behavioral Activation will be administered via Moodivate and will include the following core BA components: (1) psychoeducation, (2) development of individualized values and value-drive activities, (3) scheduling and completing activities, (4) eliciting social support to help complete difficult activities, and (5) rating daily mood and reinforcing treatment utilization. Moodivate will also be modified for a mobile environment in key ways, with the most salient being: 1) Elimination of the need for a therapist in order to reach a broad patient/consumer base that may not utilize traditional therapy resources and will combat the primary barrier to PCPs recommending psychotherapy to their patients with elevated depressive symptoms and 2) Elimination of paper forms to increase the sensitivity of BA for individuals with motivational and organizational deficits.
- Cognitive Behavioral Therapy: Moodkit (a mobile app utilizing Cognitive Behavioral Therapy techniques) will be used to administer cognitive behavioral therapy which is commonly compared to behavioral activation.
  Cognitive Behavioral Therapy (CBT) explores patterns of thinking that lead to self-destructive actions and the beliefs that direct these thoughts. CBT is an evidence-based approach for reducing depression.
Period: Overall Study
Arm/Group | Behavioral Activation | Cognitive Behavioral Therapy | Treatment as Usual
Started | 24 | 19 | 9
Completed | 22 | 18 | 9
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation | Cognitive Behavioral Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 24 | 19 | 9 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 19 | 9 | 52
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.67 (13.95) | 43.00 (13.63) | 43.11 (11.88) | 43.79 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 8 | 43
  Male | 4 | 4 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 24 | 17 | 9 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 19 | 9 | 52
Relationship Status [Count of Participants; unit: Participants]
  In a relationship | 8 | 7 | 4 | 19
  Single | 16 | 12 | 5 | 33
Education [Count of Participants; unit: Participants]
  ≤ High School Diploma | 2 | 4 | 2 | 8
  ≥ High School Diploma | 22 | 15 | 7 | 44
Annual Household Income [Count of Participants; unit: Participants]
  < $50k | 13 | 13 | 6 | 32
  ≥ $50k | 11 | 6 | 3 | 20
Employment Status [Count of Participants; unit: Participants]
  Unemployed | 3 | 2 | 2 | 7
  Employed ≥ part time | 13 | 11 | 7 | 31
  Other | 8 | 6 | 0 | 14
Phone Ownership [Count of Participants; unit: Participants]
  iPhone | 12 | 8 | 3 | 23
  Android or other smartphone | 12 | 11 | 6 | 29
Currently Taking Medication for Mental/Emotional Problems [Count of Participants; unit: Participants]
  Yes | 9 | 7 | 3 | 19
  No | 15 | 12 | 6 | 33
Current Major Depressive Episode [Count of Participants; unit: Participants]
  Yes | 17 | 14 | 6 | 37
  No | 7 | 5 | 3 | 15
Lifetime Major Depressive Episode [Count of Participants; unit: Participants]
  Yes | 23 | 17 | 9 | 49
  No | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Average Decrease of Beck Depression Inventory-II Score
Description: The BDI-II is a well-validated tool for the assessment of depressive symptoms and is our key outcome measure. For assessing weekly changes in mood, we will use the Profile of Mood States, a brief self-report scale that has demonstrated satisfactory psychometric properties. For MDD diagnosis, during the phone screening, participants will complete a shortened version of the MDD module of the Structured Clinical Interview for the DSM-IV. The scale for the Beck's Depression Inventory is 0-63 where higher scores indicate more severe depressive symptoms. Scores were analyzed as a 10 point decrease from baseline at any point in the study. For pretreatment, participants completed the BDI-II at baseline and for posttreatment, participants completed the BDI-II 8 weeks after baseline. Values were calculated by subtracting pretreatment from posttreatment and averaging across participants, within treatment condition.
Time Frame: Baseline and Week 8
Population: For pretreatment, participants completed the BDI-II at baseline and for posttreatment, participants completed the BDI-II 8 weeks after baseline.
Measure: Mean (Standard Deviation); unit: Decrease in units on scale
Arm/Group | Behavioral Activation | Cognitive Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 22 | 18 | 9
Decrease in units on scale | -12.21 (13.15) | -13.36 (11.51) | -7.75 (14.99)
Statistical Analysis 1: Comparison: Behavioral Activation vs Cognitive Behavioral Therapy vs Treatment as Usual; Test type: Other — A generalized estimating equation (GEE) model assuming a normal distribution, identity link function, and exchangeable correlation matrix was used to examine the interaction between time and treatment condition on BDI-II depressive symptoms adjusting for the main effects of baseline depressive symptoms, time, and treatment condition; p < .05, Chi-squared

2. Secondary Outcome: Client Treatment Adherence
Description: Client treatment adherence will be measured based on the activity selection and scheduling component of Moodivate.
Time Frame: Once a week for 8 weeks
Population: All participants who completed at least one follow-up assessment were included in analyses; data was only available for 21 Moodivate participants due to technical issues.
Measure: Mean (Standard Deviation); unit: Total number of Moodivate sessions compl
Arm/Group | Behavioral Activation | Cognitive Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 21 | 0 | 0
Total number of Moodivate sessions compl | 46.76 (30.10) |  |

3. Secondary Outcome: Changes Among User Feasibility and Acceptability
Description: User feasibility and acceptability will be assessed both during and following the 8 weeks of Moodivate or MoodKit treatment. During the course of Moodivate or MoodKit treatment, users will be prompted at random intervals to respond to a brief survey online assessing: 1) ease of use of the product, 2) continued desire to use the product, 3) perceived benefits of using the product, and 4) suggestions for product development/modifications for Behavioral Apptivation only). Following the 8 weeks of treatment, participants who were randomized to the Moodivate condition will attend a phone call with the Invesitgator at the Medical University of South Carolina.
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Positive and Negative Affect Schedule (PANAS)
Description: Participants completing the PANAS are asked to rate the extent to which they experienced each out of 20 emotions on a 5-point Likert Scale ranging from "very slightly" to "very much". The exact instructions may vary according to the purpose of the study: Participants may be asked how they feel right now or during longer periods of time (e.g. during the past year). Half of the presented emotion words concern negative affect (distressed, upset, guilty, ashamed, hostile, irritable, nervous, jittery, scared, afraid), the other half positive affect (interested, alert, attentive, excited, enthusiastic, inspired, proud, determined, strong, active). The PANAS is usually regarded as a reliable measure for non-clinical populations
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: EROS ( Emotion Regulation of Others and Self)
Description: Assesses strategies used to improve and worsen both one's own and others' emotions. It has two subscales. The intrinsic subscale measures emotion self-regulation using 10 items. The extrinsic subscale measures interpersonal emotion regulation using 9 items.
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Profile of Mood States (POMS)
Description: Measures affective mood states
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Behavioral Activation for Depression Scale (BADS)
Description: The Behavioral Activation for Depression Scale (BADS) can be used to track changes weekly in the behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation. It examines changes in the following areas: activation, avoidance/rumination, work/school impairment, and social impairment.
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Snaith-Hamilton Pleasure Scale (SHAPS)
Description: Assesses anhedonia a core symptom in depression
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

10. Secondary Outcome: The Addiction Severity Index (ASI) i
Description: The Addiction Severity Index (ASI) is a semi-structured interview for substance abuse assessment and treatment planning. The ASI is designed to gather valuable information about areas of a client's life that may contribute to their substance-abuse problems.
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Fagerstrom Test For Nicotine Dependence (FTND)
Description: The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Timeline Followback Method Assessment
Description: The Timeline Followback (TLFB) is a method that can be used as a clinical and research tool to obtain a variety of quantitative estimates of marijuana, cigarette, and other drug use.
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Contemplation Ladder
Description: A measure of readiness to consider smoking cessation
Time Frame: Once a week for 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Once a week for 8 weeks.
Description: The definition of adverse event and serious adverse event is consistent with the definition reported in clinicaltrials.gov.
Arm/Group | Behavioral Activation | Cognitive Behavioral Therapy | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/19 | 0/9
Other Adverse Events (participants affected / at risk) | 0/24 | 0/19 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No